CLINICAL TRIAL: NCT00222989
Title: PPI Versus Placebo in Severe Functional Heartburn
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started.
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael M Kline, Associate Professor of Clinical Medicine, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: #026020; 474200
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: GERD
Keywords: GERD; PPI; Functional heartburn
MeSH Terms: conditions — Gastroesophageal Reflux

ARMS (1):
- no label study (Other): 1
  Interventions: Drug: PPI

INTERVENTIONS:
Drug: PPI

SUMMARY:
Proton Pump Inhibitors are no better than placebo in relieving GERD symptoms in patients with functional Heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Heartburn twice a week for at least 2 years. Normal EGD and 24hr pH study.

Exclusion Criteria:

* <18yrs of age,pregnant, unable or unwilling to give consent, allergic to PPI, previous gastric or esophageal surgery, past hx of erosive GERD, unwilling or unable to stop acid suppression meds

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-10; Primary Completion 2100-12-01 (Estimated); Study Completion 2100-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in GERD controll PPI vs Placebo based on a validated GERD questionnarir. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Kline, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Keck School of Medicine, Los Angeles, California, United States